CLINICAL TRIAL: NCT00921310
Title: A Phase I/II Trial of Temsirolimus and Pemetrexed in Recurrent/Refractory Non Small Cell Lung Cancer (NSCLC)
Brief Title: Temsirolimus and Pemetrexed for Recurrent or Refractory Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawal of funding from sponsor
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0668 / 201105207
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Temsirolimus and pemetrexed for recurrent or refractory NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase I Dose Level 1 (pemetrexed + temsirolimus) (Experimental): -Dose Level 1
  * Pemetrexed 500mg/m^2 intravenous (IV) on Day 1 of each 21 day cycle
  * Temsirolimus 15 mg IV on Days 1,8 and 15 of each 21 day cycle
  Interventions: Drug: Pemetrexed; Drug: Temsirolimus
- Phase I Dose Level -1 (pemetrexed + temsirolimus) (Experimental): * Pemetrexed (375 mg/m^2) IV on Day 1 of each 21 day cycle
  * Temsirolimus (15 mg) IV on Days 1,8 and 15 of each 21 day cycle
  Interventions: Drug: Pemetrexed; Drug: Temsirolimus
- Phase 2 (pemetrexed + temsirolimus) (Experimental): * Phase 2 dose will be the maximum tolerated dose found in the Phase I portion of the study.
  * Pemetrexed (375 mg/m^2) IV on Day 1 of each 21 day cycle
  * Temsirolimus (15 mg) IV on Days 1,8 and 15 of each 21 day cycle
  Interventions: Drug: Pemetrexed; Drug: Temsirolimus

INTERVENTIONS:
Drug: Pemetrexed
  Other Names: Alimta
Drug: Temsirolimus
  Other Names: Torisel

SUMMARY:
To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of the combination of temsirolimus and pemetrexed, as well as the response rate. The starting dose (Dose Level 1) and schedule of pemetrexed will be 500 mg/m^2 given every 3 weeks and the starting dose (Dose Level 1) for temsirolimus will be 15 mg given weekly for 3 weeks, to complete 1 cycle. In subsequent cohorts, dose will be escalated or de-escalated. Enrollment to each cohort is based on toxicity experienced at that dose level.

DETAILED DESCRIPTION:
* To determine the maximum tolerated dose (MTD) of temsirolimus that could be administered weekly in combination with pemetrexed.
* To determine the dose-limiting toxicity (DLT) of temsirolimus and pemetrexed as well as other toxicities of this combination therapy.
* To describe the response rate of the combination in patients with relapsed/refractory non-small cell lung cancer (NSCLC).
* To describe phospho-Akt and phospho-S6 levels in circulating mononuclear cells before and after treatment.
* To determine the response rates in patients with NSCLC when treated with temsirolimus and pemetrexed.
* To evaluate progression-free survival in patients with NSCLC when treated with temsirolimus and pemetrexed.
* To determine the one-year survival rates in patients with NSCLC when treated with temsirolimus and pemetrexed.
* To describe phospho-Akt and phospho-S6 levels in circulating mononuclear cells before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of NSCLC.
* Patients must have non-squamous histology.
* Patients must have measurable disease (by RECIST criteria), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan.
* Patients may have failed at least one prior platinum-based therapy for NSCLC or be candidates for first-line therapy for advanced disease deemed ineligible to receive platinum-based chemotherapy in the opinion of the treating physician (e.g., Eastern Cooperative Oncology Group (ECOG) performance status of 2, age ≥ 70, chronic medical condition).
* Patients must be at least 4 weeks out from chemotherapy, biological therapy, major surgery, or any investigative therapy and must have recovered from any toxicities. Patients must be at least 2 weeks out from prior radiation therapy and must have recovered from any associated toxicities (with the exception of alopecia).
* Patients must be at least 3 weeks out from immunosuppressive therapy (except corticosteroids used as antiemetics).
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of pemetrexed in combination with temsirolimus in patients <18 years of age, children are excluded from this study.
* ECOG performance status 0-2.
* Patients must have normal organ and marrow function as defined below:

  * hemoglobin ≥9.0 g/dL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤1.5 mg/dL
  * aspartate aminotransferase (AST)(SGOT)/ alanine aminotransferase (ALT) (SGPT) ≤2.5 X institutional upper limit of normal OR ≤5 X institutional upper limit of normal if enzyme abnormalities are due to liver metastases
  * creatinine < 2.0 mg/dL AND/OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
  * serum cholesterol < 350 mg/dL
  * triglycerides < 300 mg/dL
* The effects of pemetrexed and temsirolimus on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because antifolate antineoplastic agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability of the patient (or legally authorized representative if applicable) to understand and the willingness to sign a written informed consent document.
* Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Patients who have had previous treatment with pemetrexed.
* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, clinically significant hepatic or renal disease or neuropathy greater than grade 2.
* Symptomatic brain metastases
* Presence of a third-space fluid (pleural effusion, ascites etc.) that is uncontrolled by drainage.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temsirolimus, its metabolites (including sirolimus), its components, and/or polysorbate 80, or to other agents used in the study.
* Known hypersensitivity to macrolide antibiotics.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements and with premedications of dexamethasone, folic acid and vitamin B12.
* Patients with inability to discontinue all non-steroidal anti-inflammatory drugs (NSAIDS).
* Patients taking anticonvulsant medications (Carbamezapine, phenytoin, fosphenytoin, phenobarbital).
* Patients taking anti-arrhythmic medications (amiodarone, diltiazem and quinidine).
* Patients may not be taking medications known as inhibitors of CYP3A4 (carbamezapine, phenytoin, phenobarbital, rifampin, St. John's wort). Use of inducers of CYP3A4 is discouraged but not specifically prohibited. Dexamethasone as a chronic medication is discouraged.
* Pregnant women are excluded from this study because pemetrexed is an antifolate antineoplastic drug with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pemetrexed, breastfeeding should be discontinued if the mother is treated with pemetrexed. These potential risks may also apply to other agents used in this study.
* Patients with known concomitant genetic or acquired immunosuppressive diseases are excluded. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pemetrexed and temsirolimus. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Baggstrom, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Russo F, Bearz A, Pampaloni G; Investigators of Italian Pemetrexed Monotherapy of NSCLC Group. Pemetrexed single agent chemotherapy in previously treated patients with locally advanced or metastatic non-small cell lung cancer. BMC Cancer. 2008 Jul 31;8:216. doi: 10.1186/1471-2407-8-216. PMID 18667090
- [Background] Pal SK, Figlin RA, Reckamp KL. The role of targeting mammalian target of rapamycin in lung cancer. Clin Lung Cancer. 2008 Nov;9(6):340-5. doi: 10.3816/CLC.2008.n.049. PMID 19073516
- [Background] Atkins MB, Hidalgo M, Stadler WM, Logan TF, Dutcher JP, Hudes GR, Park Y, Liou SH, Marshall B, Boni JP, Dukart G, Sherman ML. Randomized phase II study of multiple dose levels of CCI-779, a novel mammalian target of rapamycin kinase inhibitor, in patients with advanced refractory renal cell carcinoma. J Clin Oncol. 2004 Mar 1;22(5):909-18. doi: 10.1200/JCO.2004.08.185. PMID 14990647
- [Background] Rini BI. Temsirolimus, an inhibitor of mammalian target of rapamycin. Clin Cancer Res. 2008 Mar 1;14(5):1286-90. doi: 10.1158/1078-0432.CCR-07-4719. No abstract available. PMID 18316545
- [Background] Duran I, Kortmansky J, Singh D, Hirte H, Kocha W, Goss G, Le L, Oza A, Nicklee T, Ho J, Birle D, Pond GR, Arboine D, Dancey J, Aviel-Ronen S, Tsao MS, Hedley D, Siu LL. A phase II clinical and pharmacodynamic study of temsirolimus in advanced neuroendocrine carcinomas. Br J Cancer. 2006 Nov 6;95(9):1148-54. doi: 10.1038/sj.bjc.6603419. Epub 2006 Oct 10. PMID 17031397
- [Background] Peralba JM, DeGraffenried L, Friedrichs W, Fulcher L, Grunwald V, Weiss G, Hidalgo M. Pharmacodynamic Evaluation of CCI-779, an Inhibitor of mTOR, in Cancer Patients. Clin Cancer Res. 2003 Aug 1;9(8):2887-92. PMID 12912932
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 09/28/2009 and closed to participant enrollment on 12/20/2011.
Groups:
- Phase I Dose Level 1 (Pemetrexed & Temsirolimus): * Pemetrexed 500mg/m^2 intravenous (IV) on Day 1 of each 21 day cycle
  * Temsirolimus 15 mg IV on Days 1,8 and 15 of each 21 day cycle
- Phase I Dose Level -1 (Pemetrexed & Temsirolimus): * Pemetrexed (375 mg/m^2) IV on Day 1 of each 21 day cycle
  * Temsirolimus (15 mg) IV on Days 1,8 and 15 of each 21 day cycle
- Phase 2 (Pemetrexed & Temsirolimus): * Phase 2 dose will be the maximum tolerated dose found in the Phase I portion of the study.
  * Pemetrexed (375 mg/m^2) IV on Day 1 of each 21 day cycle
  * Temsirolimus (15 mg) IV on Days 1,8 and 15 of each 21 day cycle
Period: Overall Study
Arm/Group | Phase I Dose Level 1 (Pemetrexed & Temsirolimus) | Phase I Dose Level -1 (Pemetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Started | 2 | 6 | 4
Completed | 2 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I (Premetrexed & Temsirolimus): * Participants enrolled in the Phase I portion Dose Level 1 received:
    * Pemetrexed 500mg/m^2 IV on Day 1 of each 21 day cycle
    * Temsirolimus 15 mg IV on Days 1,8 and 15 of each 21 day cycle
  * Participants enrolled in the Phase I portion Dose Level -1 received:
    * Pemetrexed 375mg/m^2 IV on Day 1 of each 21 day cycle
    * Temsirolimus 15 mg IV on Days 1,8 and 15 of each 21 day cycle
- Phase 2 (Pemetrexed & Temsirolimus): -Participants enrolled in the Phase 2 portion received:
  * Pemetrexed (375 mg/m2^2) IV on Day 1 of each 21 day cycle
  * Temsirolimus (15 mg) IV on Days 1,8 and 15 of each 21 day cycle
- Total: Total of all reporting groups
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus) | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Median (Full Range); unit: years] | 58.5 [49 to 76] | 67.5 [62 to 70] | 62.5 [49 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Phase I Only: Maximum Tolerated Dose (MTD) of Pemetrexed That Could be Administered Weekly in Combination With Temsirolimus
Description: The starting dose and schedule of pemetrexed will be 500 mg/m2 given every 3 weeks and the starting dose for temsirolimus will be 15 mg given weekly for 3 weeks, to complete 1 cycle. In subsequent cohorts, dose will be escalated or de-escalated. Enrollment to each cohort is based on toxicity experienced at that dose level. The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort experience dose-limiting toxicity during the first cycle. Six patients will be enrolled at the maximum tolerated dose to ensure that no more than 2 DLTs occur at the MTD. Dose escalations will proceed until the MTD has been reached.
Time Frame: Completion of first cycle by all enrolled patients in Phase I portion of study
Measure: Number; unit: mg/m^2
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Number analyzed (Participants) | 8 | 0
mg/m^2 | 375 |

2. Primary Outcome: Phase I Only: Maximum Tolerated Dose (MTD) of Temsirolimus That Could be Administered Weekly in Combination With Pemetrexed
Description: as for outcome 1
Time Frame: Completion of first cycle by all enrolled patients in Phase I portion of study
Measure: Number; unit: mg
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Number analyzed (Participants) | 8 | 0
mg | 15 |

3. Primary Outcome: Phase I Only: Number of Participants Who Experience Dose-limiting Toxicities (DLT) of Temsirolimus and Pemetrexed
Description: DLT will be defined as occurring within the first cycle of Phase I only and will be graded according to the Common Terminology Criteria for Adverse Events v 3.0 (CTCAE)
  * Any grade 3 or higher hematologic toxicity with the exception of anemia.
  * Any grade 3 or higher non-hematologic toxicity related to study therapy (except alopecia).
  * Grade 3 or 4 pneumonitis or esophagitis.
  * Treatment delay of temsirolimus for more than 14 consecutive days due to study-related toxicity.
  * Treatment delay of pemetrexed therapy for more than 14 consecutive days because of study-related toxicity.
Time Frame: Completion of first cycle (approximately 21 days)
Measure: Number; unit: participants
Groups:
- Phase I Dose Level 1 (Premetrexed & Temsirolimus): * Pemetrexed 500mg/m^2 intravenous (IV) on Day 1 of each 21 day cycle
  * Temsirolimus 15 mg IV on Days 1,8 and 15 of each 21 day cycle
- Phase 1 Dose Level -1 (Pemetrexed & Temsirolimus): * Pemetrexed (375 mg/m^2) IV on Day 1 of each 21 day cycle
  * Temsirolimus (15 mg) IV on Days 1,8 and 15 of each 21 day cycle
Arm/Group | Phase I Dose Level 1 (Premetrexed & Temsirolimus) | Phase 1 Dose Level -1 (Pemetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Number analyzed (Participants) | 2 | 6 | 0
participants | 2 | 0 |

4. Primary Outcome: Phase I and Phase II: Overall Response Rate (Complete Response + Partial Response)
Description: * Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response.
  * Complete response (CR)-disappearance of all target lesions and disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial response (PR)-at least a 30% decrease in the sum of the longest diameter (LD) of the target lesions taking as reference the baseline sum LD
Time Frame: 2 years
Population: (4) patients in Phase 1 were not evaluable for response as they were removed from study prior to week 6 scans. One patient in Phase 2 was not evaluable due to expiring prior to week 6 scans.
Measure: Number; unit: percentage of participants
Groups:
- Phase I (Premetrexed & Temsirolimus): * Dose Level 1
    * Pemetrexed 500mg/m^2 IV on Day 1 of each 21 day cycle
    * Temsirolimus 15 mg IV on Days 1,8 and 15 of each 21 day cycle
  * Dose Level -1
    * Pemetrexed 375mg/m^2 IV on Day 1 of each 21 day cycle
    * Temsirolimus 15 mg IV on Days 1,8 and 15 of each 21 day cycle
- Phase 2 (Pemetrexed & Temsirolimus): Pemetrexed (375 mg/m^2) IV on Day 1 of each 21 day cycle
  Temsirolimus (15 mg) IV on Days 1,8 and 15 of each 21 day cycle
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Number analyzed (Participants) | 4 | 3
percentage of participants | 0 | 33.3

5. Primary Outcome: Phase I Only: Phospho-Akt Levels in Circulating Mononuclear Cells
Time Frame: Cycle 1 Day 1, one hour post completion of initial temsirolimus dose, and Cycle 1 Day 8
Population: Due to early termination of the study by withdrawal of funding by sponsor (Pfizer merged with Wyeth), the peripheral blood samples that were collected for this outcome measure were not analyzed prior to losing funding.
Groups:
- Phase 2 (Pemetrexed & Temsirolimus): Pemetrexed (375 mg/m2^2) IV on Day 1 of each 21 day cycle
  Temsirolimus (15 mg) IV on Days 1,8 and 15 of each 21 day cycle
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Phase I Only: Phospho-S6 Levels in Circulating Mononuclear Cells
Time Frame: Cycle 1 Day 1, one hour post completion of initial temsirolimus dose, and Cycle 1 Day 8
Population: as for outcome 5
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase 2 Only: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression.
Time Frame: 2 years from completion of treatment
Population: There were only (2) patients evaluable for PFS.
Measure: Number; unit: days
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Number analyzed (Participants) | 0 | 2
days
  Patient A |  | 523
  Patient B |  | 167

8. Secondary Outcome: Phase 2 Only: Survival Rate
Time Frame: 1 year after start of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Number analyzed (Participants) | 0 | 4
percentage of participants |  | 50

9. Secondary Outcome: Phase 2 Only: Phospho-Akt Levels in Circulating Mononuclear Cells
Time Frame: Cycle 1 Day 1, one hour post completion of initial temsirolimus dose, and Cycle 1 Day 8
Population: as for outcome 5
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Phase 2 Only: Phospho-S6 Levels in Circulating Mononuclear Cells Before and After Treatment
Time Frame: Cycle 1 Day 1, one hour post completion of initial temsirolimus dose, and Cycle 1 Day 8
Population: as for outcome 5
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Phase I (Premetrexed & Temsirolimus) | Phase 2 (Pemetrexed & Temsirolimus)
Serious Adverse Events (participants affected / at risk) | 2/8 | 2/4
Other Adverse Events (participants affected / at risk) | 8/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I (Premetrexed & Temsirolimus) (N=8) | Phase 2 (Pemetrexed & Temsirolimus) (N=4)
Neutrophils (ANC) (Investigations) | 1 | 0
Leukocytes (WBC) (Investigations) | 2 | 0
Platelets (Investigations) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Vascular disorders) | 2 | 1
Disease progression - death (General disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection - pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Aspiration pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I (Premetrexed & Temsirolimus) (N=8) | Phase 2 (Pemetrexed & Temsirolimus) (N=4)
ALT (Investigations) | 3 | 2
AST (Investigations) | 5 | 0
Albumin - low (Metabolism and nutrition disorders) | 3 | 4
Alkaline phosphatase (Investigations) | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 2
Bilirubin (Investigations) | 1 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0
Calcium - low (Metabolism and nutrition disorders) | 3 | 1
Chest pain (Cardiac disorders) | 1 | 0
Chloesterol - high (Investigations) | 0 | 2
Confusion (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Creatinine (Investigations) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Edema (General disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Fatigue (General disorders) | 3 | 3
Fever (General disorders) | 0 | 2
Glucose - high (Metabolism and nutrition disorders) | 5 | 2
Hand pain (Investigations) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Hemoglobin (Blood and lymphatic system disorders) | 7 | 4
Hot flashes (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INR (Investigations) | 1 | 0
Infusion reaction (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 3
Leukocytes (WBC) (Investigations) | 6 | 3
Lymphopenia (Investigations) | 8 | 4
Magnesium - low (Metabolism and nutrition disorders) | 1 | 0
Mood alteration - anxiety (Psychiatric disorders) | 0 | 1
Mood alteration - depression (Psychiatric disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 3
Neutrophils (ANC) (Investigations) | 3 | 3
Pain NOS (General disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Phosphorus - low (Metabolism and nutrition disorders) | 2 | 1
Platelets (Investigations) | 5 | 4
Potassium - high (Metabolism and nutrition disorders) | 2 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sensory neuropathy (Nervous system disorders) | 0 | 1
Skin breakdown/decubitous ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Sodium - low (Metabolism and nutrition disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Sweating (General disorders) | 0 | 1
Throat pain (Investigations) | 1 | 0
Triglycerides - high (Investigations) | 1 | 1
Upper respiratory infection (Infections and infestations) | 3 | 0
Viral flare (herpes) (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Watery eyes (Eye disorders) | 1 | 1
Weight loss (Investigations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes